CLINICAL TRIAL: NCT07358637
Title: Artificial Intelligence Enhanced Optical Coherence Tomography (AI-OCT) Imaging for Pre-surgical Margin Detection of Basal Cell Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David M. Ozog, Principal Investigator, Henry Ford Health System
Other Study IDs: 18605
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Basal Cell Carcinoma of Skin
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Diagnostic Test: AI-OCT — Optical Coherence Tomography augmented by artificial intelligence software

SUMMARY:
Basal cell carcinomas (BCCs) are the most common human malignancy, affecting about 2 million Americans each year. Mohs micrographic surgery (MMS) removes tissue by sequential excision. Costs for MMS could be reduced if the number of necessary excision stages were decreased by a more accurate initial tumor margin assessment.

The goal of this observational study is to learn if Optical Coherence Tomography (OCT) used in conjunction with artificial intelligence algorithms is accurate in the detection of superficial BCC margins prior to MMS. This study also aims to determine if AI-OCT guided margin delineation can reduce the number of stages in MMS.

Researchers will first focus on validating AI-OCT as a method for accurately detecting BCCs. A follow-up study would then address the guided pre-surgical margin delineation.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, ages 18 or older
* at least one biopsy proven superficial or nodular BCC
* willingness to have photographs taken of the treatment area
* ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* infiltrative, micronodular, or morpheaform BCC
* pregnant women
* subjects not willing to have a biopsy taken from the treatment area
* subjects with herpes simplex virus infection in the treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with biopsy-confirmed BCC who are scheduled to receive Mohs micrographic surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Validation of AI-OCT as an accurate method for detecting basal cell carcinomas | 2 years